CLINICAL TRIAL: NCT03732534
Title: Open-Label Rollover Study for Continuing NBI-98854 Administration for the Treatment of Pediatric Subjects With Tourette Syndrome
Brief Title: Rollover Study for Continuing NBI-98854 Administration in Pediatric Subjects With Tourette Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped early due to investigational drug not meeting primary endpoint in the main study T-Force GOLD (NBI-98854-TS2003); no safety concerns identified.
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-98854-TS2007
Record Dates: First submitted 2018-11-05; First posted 2018-11-06 (Actual); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NBI-98854 (Experimental): NBI-98854 administered once daily for up to 96 weeks
  Interventions: Drug: NBI-98854

INTERVENTIONS:
Drug: NBI-98854 — vesicular monoamine transporter 2 (VMAT2) inhibitor
  Other Names: Valbenazine

SUMMARY:
This is an open-label, rollover study to collect long-term safety, tolerability, and investigator- and participant-reported pharmacodynamic (PD) data after chronic administration of NBI-98854 in pediatric participants with Tourette Syndrome (TS), as well as to provide open-label access to NBI-98854 for the treatment of TS for pediatric participants who have taken part in a Phase 2 NBI-98854 study.

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of Tourette Syndrome (TS)
2. Have participated in the NBI-98854-TS2004 or NBI 98854-TS2005 Phase 2 studies
3. If using maintenance medication(s) for TS and/or TS spectrum diagnoses (e.g. obsessive-compulsive disorder [OCD], Attention-Deficit Hyperactivity Disorder [ADHD]), be on stable doses
4. Be in good general health
5. Subjects of childbearing potential who do not practice total abstinence must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment and follow-up periods of the study

Exclusion Criteria:

1. Have an active, clinically significant unstable medical condition within 1 month before screening
2. Have a known history of long QT syndrome or cardiac arrhythmia
3. Have a known history of neuroleptic malignant syndrome
4. Have a cancer diagnosis within 3 years prior to screening (some exceptions allowed)
5. Have an allergy, hypersensitivity, or intolerance to VMAT2 inhibitors
6. Have a blood loss ≥250 mL or donated blood within 56 days, or donated plasma within 7 days, before the start of the study
7. Have a known history of substance dependence, substance (drug) or alcohol abuse within 3 months before the start of the study
8. Have a significant risk of suicidal or violent behavior
9. Have received an investigational drug within 30 days before the start of the study or plan to use an investigational drug (other than NBI-98854) during the study
10. Are currently participating in another NBI-98854 clinical study
11. Are pregnant (for females)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (10):
- United States (9):
  - Neurocrine Clinical Site, Anaheim, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, Gulf Breeze, Florida
  - Neurocrine Clinical Site, Hialeah, Florida
  - Neurocrine Clinical Site, Chicago, Illinois
  - Neurocrine Clinical Site, Naperville, Illinois
  - Neurocrine Clinical Site, Lincoln, Nebraska
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, Houston, Texas
- Neurocrine Clinical Site, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 240 participants who completed the Phase 2 Study NBI-98854-TS2004 or were to be dosed for at least 16 weeks in Phase 2 Study NBI-98854-TS2005 were planned for this study. However, only 6 participants were enrolled and received study drug because the study was terminated early by the Sponsor.
Groups:
- Valbenazine: Participants received valbenazine once daily for up to 96 weeks. The starting dose was 20 mg for participants <50 kg at baseline and 40 mg for participants ≥50 kg at baseline, and could be escalated in increments of 20 mg every 2 weeks to a maximum of 60 mg for participants <50 kg and 80 mg for participants ≥50 kg to achieve an optimal dose of valbenazine for each participant.
Period: Overall Study
Arm/Group | Valbenazine
Started | 6
Completed | 0
Not Completed | 6
Not completed — Study terminated by Sponsor | 6

BASELINE CHARACTERISTICS:
Arm/Group | Valbenazine
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE is an adverse event not present prior to the initiation of study drug dosing, or is an already present event that worsens either in intensity or frequency following the initiation of study drug dosing.
Time Frame: Up to 16 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Valbenazine
Number analyzed (Participants) | 6
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Arm/Group | Valbenazine
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine (N=6)
Somnolence (Nervous system disorders) | 2
Nasopharyngitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT03732534/Prot_SAP_000.pdf